CLINICAL TRIAL: NCT00249912
Title: A Double-Blind, Randomized Study to Evaluate the Efficacy and Safety of Lapaquistat Acetate 50 mg, 100 mg or Placebo When Coadministered With Rosuvastatin 10 mg or 20 mg in Subjects With Primary Hypercholesterolemia
Brief Title: Efficacy of Lapaquistat Acetate Alone or Combined With Rosuvastatin in Subjects With Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-05-TL-475-022; U1111-1122-8106 (Registry Identifier: WHO)
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Hypercholesterolemia
Keywords: Hyperlipidemia; Drug Therapy
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias | interventions — 1-((1-(3-acetoxy-2,2-dimethylpropyl)-7-chloro-5-(2,3-dimethoxyphenyl)-2-oxo-1,2,3,5-tetrahydro-4,1-benzoxazepin-3-yl)acetyl)piperidine-4-acetic acid; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lapaquistat Acetate 50 mg QD + Rosuvastatin (Experimental)
  Interventions: Drug: Lapaquistat acetate and rosuvastatin
- Lapaquistat Acetate 100 mg QD + Rosuvastatin (Experimental)
  Interventions: Drug: Lapaquistat acetate and rosuvastatin
- Rosuvastatin (Active Comparator)
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Lapaquistat acetate and rosuvastatin — Lapaquistat acetate 50 mg, tablets, orally, once daily and stable Rosuvastatin therapy (10 or 20 mg) for up to 24 weeks.
  Other Names: TAK-475; Crestor
  Arms: Lapaquistat Acetate 50 mg QD + Rosuvastatin
Drug: Lapaquistat acetate and rosuvastatin — Lapaquistat acetate 100 mg, tablets, orally, once daily and stable Rosuvastatin therapy (10 or 20 mg) for up to 24 weeks.
  Other Names: TAK-475; Crestor
  Arms: Lapaquistat Acetate 100 mg QD + Rosuvastatin
Drug: Rosuvastatin — Lapaquistat acetate placebo-matching tablets, orally, once daily and stable Rosuvastatin therapy (10 or 20 mg) for up to 24 weeks.
  Other Names: Crestor
  Arms: Rosuvastatin

SUMMARY:
The purpose of this study is to evaluate lapaquistat acetate, once daily (QD), taken alone or with rosuvastatin on cholesterol levels in treating patients with elevated cholesterol.

DETAILED DESCRIPTION:
Elevated plasma cholesterol (hypercholesterolemia) and various other plasma lipid imbalances (dyslipidemias) are major risk factors for coronary heart disease. Patients with hypercholesterolemia have elevated low-density lipoprotein cholesterol, which leads to atherosclerotic deposition of cholesterol in the arterial walls. As identified by the National Cholesterol Education Program Adult Treatment Panel III, lowering the low-density lipoprotein cholesterol plasma concentration effectively reduces cardiovascular morbidity and mortality and is essential for the prevention and management of coronary heart disease.

Currently, 3-hydroxy-3-methylglutaryl-coenzyme A reductase inhibitors (statins) are the first-line monotherapies prescribed to reduce low-density lipoprotein cholesterol, after diet and therapeutic lifestyle change. However, low doses of statins often fail to produce the ATP III-recommended levels of low-density lipoprotein cholesterol reduction, making it necessary to increase the dose or add an additional treatment. Dose increases of statins in turn may result in decreased tolerability and potential safety concerns which contribute to the high discontinuation rates of statins and their prescription at low, and often ineffective, doses.

The purpose of this study is to determine whether administration of lapaquistat acetate co-administered with rosuvastatin will be more efficacious in lowering low-density lipoprotein cholesterol, compared to lapaquistat or rosuvastatin alone. Total participation time in this study is anticipated to be 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Woman of childbearing potential can not to be pregnant, lactating, not planning on becoming pregnant, and agree to use acceptable forms of contraception throughout the course of the study.
* Prior to Randomization, has a low-density lipoprotein cholesterol level mean greater than or equal to 3.37 mmol/L and less than or equal to 5.70 mmol/L.
* Prior to Randomization, has a mean triglyceride level less than or equal to 4.52 mmol/L (400 mg/dL).
* Has clinical laboratory evaluations including clinical chemistry, hematology, and urinalysis within the defined reference range.
* Participant is taking a stable dose of rosuvastatin (10 or 20 mg) for at least 4 weeks prior to Screening.

Exclusion Criteria:

* Has an alanine aminotransferase or aspartate aminotransferase level of greater than 1.5 times the upper limit of normal, active liver disease or jaundice.
* Has a serum creatinine of greater than 133 μmol/L.
* Has a creatine kinase greater than 3 times the upper limit of normal.
* Has type 1 or 2 diabetes mellitus.
* Has a previous history of cancer that had been in remission for less than 5 years prior to the first dose of study medication.
* Has an endocrine disorder, such as Cushing syndrome, hyperthyroidism, or inappropriately treated hypothyroidism, affecting lipid metabolism.
* Has a history of myocardial infarction, angina pectoris, transient ischemic attacks, cerebrovascular accident, peripheral vascular disease, abdominal aortic aneurysm, coronary revascularization or multiple factors that conferred a 10-year risk for coronary heart disease greater than 20% based on Framingham risk scoring.
* Has a positive hepatitis B surface antigen, or antibody to hepatitis C virus, as determined by medical history and/or subject's verbal report.
* Has a positive human immunodeficiency virus status or was taking antiretroviral medications, as determined by medical history.
* Has exposure to lapaquistat acetate in other studies, was participating in another investigational study, or had participated in an investigational study within the past 30 days or, for drugs with a long half-life, within a period of less than 5 times the drug's half-life.
* The subject had a known hypersensitivity or history of adverse reaction rosuvastatin.
* Has a history or presence of clinically significant food allergy that would prevent adherence to the recommended diet.
* Has a known heterozygous or homozygous familial hypercholesterolemia or known Type III hyperlipoproteinemia (familial dysbetalipoproteinemia).
* Has fibromyalgia, myopathy, rhabdomyolysis or unexplained muscle pain.
* Has uncontrolled hypertension
* Has inflammatory bowel disease, any other malabsorption syndrome, or had gastric bypass or any other surgical procedure for weight loss.
* Is unwilling or unable, in the opinion of the investigator, to comply with the protocol or scheduled appointments.
* Has a history of drug abuse or a history of alcohol abuse within the past 2 years.
* Has any other serious disease or condition that might reduced life expectancy, impaired successful management according to the protocol, or make the participant an unsuitable candidate to receive study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2005-10; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Low Density Lipoprotein cholesterol | Week 24 or Final Visit

SECONDARY OUTCOMES:
Adverse Events | Weeks: 2, 4, 8, 12, 16, 20, and 24 or Final Visit
Physical Examination | Week 24 or Final Visit
Safety Laboratory Tests | Weeks: 2, 4, 8, 12, 16, 20, and 24 or Final Visit
12- lead Electrocardiogram assessments | Week 24 or Final Visit
Best Corrected Visual Acuity results | Week 24 or Final Visit
Vital Signs | Weeks: 2, 4, 8, 12, 16, 20, and 24 or Final Visit
Change from Baseline in Triglycerides | Week 24 or Final Visit
Change from Baseline in Total Cholesterol | Week 24 or Final Visit
Change from Baseline in High Density Lipoprotein cholesterol | Week 24 or Final Visit
Change from Baseline in Very Low Density Lipoprotein cholesterol | Week 24 or Final Visit
Change from Baseline in apolipoprotein A1 | Week 24 or Final Visit
Change from Baseline in apolipoprotein B | Week 24 or Final Visit
Change from Baseline in non- High Density Lipoprotein cholesterol | Week 24 or Final Visit
Change from Baseline in the ratio of Low Density Lipoprotein cholesterol/High Density | Week 24 or Final Visit
Change from Baseline in the ratio of Total Cholesterol/High Density Lipoprotein cholesterol | Week 24 or Final Visit
Change from Baseline in the ratio of apolipoprotein A1/apolipoprotein B | Week 24 or Final Visit
Change from Baseline in high-sensitivity C-reactive protein | Week 24 or Final Visit
Percentage of subjects who achieve Low Density Lipoprotein cholesterol concentrations less than 1.81 mmol/L (70 mg/dL) | Week 24 or Final Visit
Percentage of subjects who achieve Low Density Lipoprotein cholesterol concentrations less than 2.59 mmol/L (100 mg/dL) | Week 24 or Final Visit
Percentage of subjects who achieve Low Density Lipoprotein cholesterol concentrations less than 3.37 mmol/L (130 mg/dL) | Week 24 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (92):
- United States (82):
  - Birmingham, Alabama
  - Haleyville, Alabama
  - Mobile, Alabama
  - Scottsdale, Arizona
  - Long Beach, California
  - Mission Viejo, California
  - Orange, California
  - Redondo Beach, California
  - Rolling Hills Estates, California
  - San Diego, California
  - Torrance, California
  - Tustin, California
  - Avon, Connecticut
  - Bristol, Connecticut
  - DeLand, Florida
  - Fort Lauderdale, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Naples, Florida
  - Ocala, Florida
  - Pembroke Pines, Florida
  - Plantation, Florida
  - Hayden Lake, Idaho
  - Meridian, Idaho
  - Arlington Heights, Illinois
  - Aurora, Illinois
  - Chicago, Illinois
  - Peoria, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Kansas City, Kansas
  - Witchita, Kansas
  - Louisville, Kentucky
  - Thibodaux, Louisiana
  - Auburn, Maine
  - Haverhill, Massachusetts
  - Benzonia, Michigan
  - Detroit, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Missoula, Montana
  - Concord, New Hampshire
  - West Seneca, New York
  - Raleigh, North Carolina
  - Statesville, North Carolina
  - Winstom-Salem, North Carolina
  - Grand Forks, North Dakota
  - Akron, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Kettering, Ohio
  - Tulsa, Oklahoma
  - Eugene, Oregon
  - Portland, Oregon
  - Lansdale, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Scotland, Pennsylvania
  - Cranston, Rhode Island
  - Anderson, South Carolina
  - Bristol, Tennessee
  - Cordova, Tennessee
  - Kingsport, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - McKinney, Texas
  - Midland, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Burke, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Weber City, Virginia
  - Bellevue, Washington
  - Burien, Washington
  - Edmonds, Washington
  - Seattle, Washington
  - Spokane, Washington
- Canada (10):
  - Calgary, Alberta
  - Portage la Prairie, Manitoba
  - London, Ontario
  - Oakville, Ontario
  - Oshawa, Ontario
  - Thornhill, Ontario
  - Toronto, Ontario
  - Chicoutimi, Quebec
  - Saint-Jérôme, Quebec
  - Ste-Foy, Quebec

REFERENCES:
- [Result] Stein EA, Bays H, O'Brien D, Pedicano J, Piper E, Spezzi A. Lapaquistat acetate: development of a squalene synthase inhibitor for the treatment of hypercholesterolemia. Circulation. 2011 May 10;123(18):1974-85. doi: 10.1161/CIRCULATIONAHA.110.975284. Epub 2011 Apr 25. PMID 21518985